CLINICAL TRIAL: NCT00272116
Title: Effect of Zinc and Vitamin A Supplementation on Diarrhea, Physical Growth and Immune Response in Malnourished Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Society for Applied Studies (Other)
Collaborators: European Commission (Other); World Health Organization (Other); Norwegian Council of Universities' Committee for Development Research and Education (Other)
Responsible Party: Principal Investigator, NBhandari, Director, Society for Applied Studies
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ERB3514PL950371; IC18-CT96-0045
Record Dates: First submitted 2006-01-02; First posted 2006-01-04 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-04

CONDITIONS: Diarrhea; Pneumonia; Acute Respiratory Tract Infection
Keywords: zinc; diarrhea; severe diarrhea; recurrent diarrhea; acute lower respiratory infection; pneumonia
MeSH Terms: conditions — Diarrhea; Pneumonia | interventions — Zinc; Vitamin A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 10 mg/day of elemental zinc as zinc gluconate to infants and 20 mg/day to older children and Vitamin A 100,000 IU to infants and 200,000 IU to older children
  Interventions: Drug: Zinc and vitamin A single dose at enrollment
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo and vitamin A single dose at enrollment

INTERVENTIONS:
Drug: Zinc and vitamin A single dose at enrollment — 10 mg/day of elemental zinc as zinc gluconate to infants and 20 mg/day to older children
  Arms: 1
Drug: Placebo and vitamin A single dose at enrollment — Placebo was plain glucose. Vitamin A 100,000 IU to infants and 200,000 IU to older children
  Arms: 2

SUMMARY:
Zinc deficiency is common in developing country children, as food intakes are often low, foods from animal sources are infrequently used, the bioavailability of zinc from staple cereal-based diets is limited and zinc losses occur during recurring diarrheal illnesses. Zinc deficiency is associated with impairment in immunological and other defenses against infection and increased rates of serious infections. Due to limitations in currently used biochemical markers, supplementation trials in populations likely to be deficient provide a reliable means of assessing health consequences of zinc deficiency.

A significantly lower incidence and prevalence of diarrhea has been observed in zinc supplemented developing country children in several placebo-controlled trials. The effect of routine zinc supplementation on lower respiratory tract infection is still unclear. We, therefore, evaluated the impact of daily zinc supplementation in a representative sample of children aged 6 to 30 months enrolled from a New Delhi slum area, with a sample size sufficient to determine the impact on the incidence of severe diarrhea and acute lower respiratory infection.

DETAILED DESCRIPTION:
Diarrheal disease is a major cause of child mortality in developing countries. Currently, the management of diarrhea focuses on oral rehydration therapy in acute diarrhea. However, acute diarrhea accounts for only 1/3 of the diarrhea-related deaths, the majority of the remaining being caused by persistent diarrhea. Currently persistent diarrhea treatment is complex, not yet adapted to community settings and, hence, has only a marginal impact on diarrheal mortality. A major challenge is to develop and implement cost-effective community-based interventions that can be applied to children with diarrhea to prevent persistence.

The trial was implemented in the urban slum of Dakshinpuri comprising 15,000 dwellings and a population of about 75,000. Recent data from a neighboring community indicated that childhood malnutrition, zinc deficiency, diarrhea and lower respiratory tract infection were common. Children aged 6 to 30 months were identified through a door-to-door survey. Enrollment required that the parents give informed consent and that families did not intend to emigrate. Eligible children were individually randomized by a simple randomization scheme in blocks of 8 generated by a person at Statens Serum Institut, Denmark. The zinc and placebo syrups were prepared and packaged in unbreakable bottles by GK Pharma Aps (Koge, Denmark( and labeled with unique child number according to the randomization scheme. The zinc and placebo syrups were similar in appearance, taste and packaging.

The enrolled children were randomized to receive zinc gluconate (10 mg elemental zinc/day to infants and 20 mg/day to older children) or placebo daily for a period of 4 months. All included subjects were given a massive dose of vitamin A at enrollment in addition to zinc or placebo. A field attendant administered the syrup daily at home for 4 months except on Sundays, when the mother was asked to administer it. One bottle containing 250 mL was kept in the child's home and replaced monthly.

Field workers visited households every seventh day during the 4-month follow-up period. At each visit, information was obtained for the previous 7 days on history of fever, number and consistency of stools. If the child had diarrhea or vomiting, dehydration was assessed. Information was also obtained on cough, lower chest indrawing and on their illness characteristics and whether treatment was sought in the previous 7 days. Intervention impact was assessed on physician-diagnosed acute lower respiratory tract infections and pneumonia.

Blood was collected at baseline in all children to measure micronutrient status. Cognitive development was measured at baseline and end study using Bayelys Scales of Infant Development version II.

ELIGIBILITY:
Inclusion Criteria:

* Children in the age group 6-30 months
* Either sex

Exclusion Criteria:

* Refused consent
* Likely to move out of study area within the next four months
* Urgent admission to hospital on the enrollment day
* Had received massive dose of vitamin A within the two months before enrollment

Ages: 6 Months to 30 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2482 (Actual)
Dates: Start 1998-02; Primary Completion 2000-02 (Actual); Study Completion 2000-09 (Actual)

PRIMARY OUTCOMES:
- To measure the impact of zinc and vitamin A on the duration of diarrheal illness | Weekly home visits for 6 months

SECONDARY OUTCOMES:
- To measure the impact of supplementation on the outcome of acute diarrhea, particularly on the risk of persistence | Weekly home visits for 6 months
- To measure the impact of supplementation on immune response to parenteral live measles vaccine and oral live tetravalent rotavirus vaccine | At baseline and end study
To measure the impact of zinc and vitamin A on cognitive development | 6 months
  Measure the efficacy of daily zinc administration on cognitive development in children 12 to 18 months of age.
-To measure the prevalence of zinc, copper, folate, vitamin B12, vitamin D, vitamin A and vitamin E deficiencies in the included children | 6 months
  From the plasma specimen collected at baseline, measure the concentration of various nutrients to estimate the prevalences of deficiency of these.
-To measure the association between nutrient status at baseline (including micronutrient status) and subsequent diarrheal and respiratory illnesses | 6 months
  Measure to what extent plasma levels of zinc, copper, folate, vitamin B12, vitamin D, vitamin A, and vitamin E predicts infections over the subsequent 4 months.
-To measure the association between nutrient status at baseline (including micronutrient status) and cognitive development. | 6 months
  We will measure to what extent, deficiencies of micronutrients predicts cognitive development in children 12 to 18 months of age.
-To measure whether or not deficiencies of selected micronutrients modifies the effect of zinc on diarrhea or pneumonia | 6 months
  From the analyses of vitamins and minerals in plasma, we will measure to what extent deficiencies of these modifies the effect of zinc on pneumonia and diarrhea.

CONTACTS AND LOCATIONS:
Overall Officials: Maharaj K Bhan, MD, Principal Investigator — All India Institute of Medical Sciences; Nita Bhandari, PhD, Principal Investigator — Society for Applied Studies, New Delhi
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Result] Bhandari N, Bahl R, Taneja S, Strand T, Molbak K, Ulvik RJ, Sommerfelt H, Bhan MK. Effect of routine zinc supplementation on pneumonia in children aged 6 months to 3 years: randomised controlled trial in an urban slum. BMJ. 2002 Jun 8;324(7350):1358. doi: 10.1136/bmj.324.7350.1358. PMID 12052800
- [Result] Bhandari N, Bahl R, Taneja S, Strand T, Molbak K, Ulvik RJ, Sommerfelt H, Bhan MK. Substantial reduction in severe diarrheal morbidity by daily zinc supplementation in young north Indian children. Pediatrics. 2002 Jun;109(6):e86. doi: 10.1542/peds.109.6.e86. PMID 12042580
- [Derived] Strand TA, Taneja S, Ueland PM, Refsum H, Bahl R, Schneede J, Sommerfelt H, Bhandari N. Cobalamin and folate status predicts mental development scores in North Indian children 12-18 mo of age. Am J Clin Nutr. 2013 Feb;97(2):310-7. doi: 10.3945/ajcn.111.032268. Epub 2013 Jan 2. PMID 23283502
- [Derived] Manger MS, Taneja S, Strand TA, Ueland PM, Refsum H, Schneede J, Nygard O, Sommerfelt H, Bhandari N. Poor folate status predicts persistent diarrhea in 6- to 30-month-old north Indian children. J Nutr. 2011 Dec;141(12):2226-32. doi: 10.3945/jn.111.144220. Epub 2011 Oct 19. PMID 22013199
- [Derived] Manger MS, Strand TA, Taneja S, Refsum H, Ueland PM, Nygard O, Schneede J, Sommerfelt H, Bhandari N. Cobalamin status modifies the effect of zinc supplementation on the incidence of prolonged diarrhea in 6- to 30-month-old north Indian children. J Nutr. 2011 Jun;141(6):1108-13. doi: 10.3945/jn.110.127415. Epub 2011 Apr 27. PMID 21525251
- [Derived] Taneja S, Strand TA, Sommerfelt H, Bahl R, Bhandari N. Zinc supplementation for four months does not affect growth in young north Indian children. J Nutr. 2010 Mar;140(3):630-4. doi: 10.3945/jn.109.115766. Epub 2010 Jan 27. PMID 20107146